CLINICAL TRIAL: NCT05888779
Title: Beverages for Thought: Exploring the Relationship Between Blood Glucose and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GFHNRC156
Record Dates: First submitted 2023-05-04; First posted 2023-06-05 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Overweight
Keywords: Healthy Weight
MeSH Terms: conditions — Overweight | interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beverage One (Milk) (Experimental): Participants will consume milk prior to completing a novel cognitive assessment on paper.
  Interventions: Other: Beverage One (Milk)
- Beverage Two (Juice) (Experimental): Participants will consume a fruit drink prior to completing a novel cognitive assessment on paper.
  Interventions: Other: Beverage Two (Juice)

INTERVENTIONS:
Other: Beverage One (Milk) — Participant will consume beverage one (milk) and complete novel cognitive assessment questionnaire on paper.
  Arms: Beverage One (Milk)
Other: Beverage Two (Juice) — Participant will consume beverage two (fruit drink) and complete novel cognitive assessment questionnaire on paper.
  Arms: Beverage Two (Juice)

SUMMARY:
The objective of this study is to conduct novel research on the relationship between blood sugar and cognition.

DETAILED DESCRIPTION:
This study is an acute parallel study design with one intervention visit needed per participant. There are 2 groups and 80 participants will be randomized into each group. Following the consent process, participants in each group will be seated individually in quiet rooms, with written instructions, several magazines, and a mini-fridge with beverages containing 110-120 kcals/8 fl oz. Participants will be provided instructions for the study, stating, "The study we are conducting explores the relationship between blood glucose and cognitive abilities. After consuming food or drink, your body regulates your blood glucose. Physical exertion can also affect blood glucose. Therefore, we ask that you relax in this space for 10-15 minutes. You can read the provided magazines during this time. Drinking a beverage will bring your body's blood glucose into the right phase for our questionnaires. In the fridge are some beverages, and we ask that you drink something."

After 10-15 minutes, participants will be given a cognitive test (a questionnaire on paper) and asked to complete as much of it as they can within 5 minutes. Then, moving to a separate area, weight and height measurements will be taken.

ELIGIBILITY:
Inclusion Criteria:

* No food allergies or food intolerances
* Healthy (no chronic disease) as determined by online questionnaire
* Non-pregnant and non-lactating
* Not currently dieting or planning to follow a special diet
* Minimal restricted eating practices

Exclusion Criteria:

* Pregnant or lactating
* Currently dieting or planning to follow a special diet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Written cognitive task results from novel cognitive assessment questionnaire. | 10 minutes post beverage ingestion
  Results of cognitive task after consuming a study beverage (milk or fruit-flavored drink). More questions answered correctly results in a higher score. The assessment has a total of 10 questions, and participants will be asked to complete as much of this assessment as they can within a 5 minute timeframe.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Hess, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2025-04-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT05888779/ICF_000.pdf